CLINICAL TRIAL: NCT03461575
Title: A Multicenter, Randomized, Double Blind, Restasis®-Controlled Non-inferiority, Moisview® Eye Drops-controlled Superiority, Phase III Study to Evaluate the Efficacy and Safety of HU007 Eye Drops in Patients With Dry Eye Syndrome
Brief Title: Efficacy and Safety of HU007 Eye Drops in Patients With Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HU-007_P3
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2018-04

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HU007 (Experimental): Cyclosporine 0.02%, trehalose 3%
  1 drop b.i.d at 12hr interval for 12 weeks
  Interventions: Drug: HU007
- Restasis (Active Comparator): Cyclosporine 0.05%
  1 drop b.i.d at 12hr interval for 12 weeks
  Interventions: Drug: Restasis
- Moisview (Active Comparator): trehalose 3%
  1 drop b.i.d at 12hr interval for 12 weeks
  Interventions: Drug: Moisview

INTERVENTIONS:
Drug: HU007 — cyclosporine 0.02%, trehalose 3%
  Arms: HU007
Drug: Restasis — cyclosporine 0.05%
  Arms: Restasis
Drug: Moisview — trehalose 3%
  Arms: Moisview

SUMMARY:
A multicenter, Randomized, Double blind, Restasis®-controlled Non-inferiority, Moisview® Eye Drops-controlled Superiority, Phase III Study to Evaluate the Efficacy and Safety of HU007 Eye Drops in Patients with Dry Eye Syndrome

ELIGIBILITY:
Inclusion Criteria:

* age over 19
* Corneal staining score(Oxford grading) ≥ 2 or Schirmer test ≤ 10mm/5min (If Schirmer test = 0mm/5min, Nasal stimulation schirmer test ≥ 3mm/5min)
* Volunteer who went through menopause more than 1 years ago before screening or has surgical menopause or who has negative result of pregnancy test or use effective contraception

Exclusion Criteria:

* The patients with systemic or ocular disorders affected the test result
* Current or recent patients used dry eye syndrome medications (topical or systemic) that may affect the status
* Being treated with systemic steroid
* Wearing contact lenses within 72 hr of screening visit
* Pregnancy or Breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
change from Baseline in Corneal staining(Oxford grading) score | Week 12

SECONDARY OUTCOMES:
change from Baseline in Corneal staining(Oxford grading) score | Week 4,8
change from Baseline of Conjunctival staining(Oxford grading) score | Week 4,8,12
change from Baseline of Strip meniscometry assessment | Week 4,8,12
change from Baseline of Tear film break-up time | Week 4,8,12
change from Baseline of Standard patient evaluation of eye dryness questionnaire | Week 4,8,12
arrival time of 100% clearence in Corneal staining test | Week 0-12
The number of total rescue drug usage | Week 0-12

CONTACTS AND LOCATIONS:
Overall Officials: Namsick Kim, Study Director — Huons Co., Ltd.; Choun-Ki Joo, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul ST.Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No